CLINICAL TRIAL: NCT01980797
Title: International Bicuspid Aortic Valve Consortium (BAVCon)
Acronym: BAVCon
Status: Active, not recruiting | Type: Observational
Sponsor: Boston University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: H-39760; 1R21HL150373-01 (NIH)
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Bicuspid Aortic Valve Disease; Thoracic Aortic Disease in Patients With a Bicuspid Aortic Valve
Keywords: Bicuspid aortic valve disease; Thoracic aortic disease; Genetics; Echocardiography; Cardiac CT; Cardiac MRI
MeSH Terms: conditions — Bicuspid Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — We are collecting DNA from either saliva or blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bicuspid aortic valve disease: Group/Cohort Label - Bicuspid aortic valve
  Group/Cohort Description -
  * Patients diagnosed with bicuspid aortic valve
  * All ages ≥8 years
  * Able to provide fully informed consent
- Tricuspid aortic valve control patients: Group/Cohort Label - Tricuspid aortic valve control patients
  Group/Cohort Description -Control patients will come from approximately matched patients without an identified bicuspid aortic valve who are trace, gender and geographically matched.
  * Patients not diagnosed with bicuspid aortic valve
  * All ages ≥8 years
  * Able to provide fully informed consent

SUMMARY:
Bicuspid aortic valve (BAV) disease is the most frequent congenital cardiac malformation, occurring in 0.5-1.2% of the US population. In young adults, it is generally a benign abnormality; but in older adults it is associated with thoracic aortic aneurysm or dissection in 20-30% of those with BAV. BAV is strongly associated with early development of aortic valve calcification or incompetence in >50% of BAV patients, and accounts for ~40% of the >30,000 aortic valve replacements (AVR) performed in the US each year. Yet, we know little of the etiology, cellular events and modifiers of progression of BAV to calcific aortic valve disease and we still do not understand the genetic cause(s) of BAV despite evidence for its high heritability.

The Specific Aims of this study are:

1. To identify the genetic causes of bicuspid aortic valve disease and its associated thoracic aortic disease.
2. To identify potential pathways to predict the clinical course of BAV disease and for treating human BAV disease.

To achieve these aims, we have created the International Bicuspid Aortic Valve Consortium (BAVCon), a consortium of institutions with cohorts of BAV patients and the expertise to fulfill the performance of these aims.

DETAILED DESCRIPTION:
The International Bicuspid Aortic Valve Consortium (BAVCon) Registry is the data collection arm of the International Bicuspid Aortic Valve Consortium, a 16 institution international consortium of investigators with interests in the genetics, molecular biology, imaging, surgery and natural history of bicuspid aortic valve disease.

The BAVCon Registry is a longitudinal cohort study, which is observational by design. The cohort will consist of patients with BAV. Consideration will be given to eventual inclusion of a disease-free control or comparison group. The study will compare genetic risk factors, cross-sectional and longitudinal data on risk factors related to the diagnosis, treatment and outcomes among groups of enrolled patients. As part of the natural course of clinical care, the patients and their physicians will determine the approach to treatment and the study will record the observed related outcomes. The study will not attempt to interfere with the outcomes through any type of planned intervention; therefore, there are no anticipated adverse events as a result of study participation.

Study Design

The Registry is designed to capture information on patients with bicuspid aortic valve disease. The BAVCon Registry population will be comprised of patients from sixteen BAVCon Clinical Centers. The participating BAVCon Clinical Centers are:

* Boston University School of Medicine, Boston (Dr. Simon Body, Consortium PI)
* GenTAC Consortium (Dr. Kim Eagle, PI)
* Hospital Vall d'Hebron, Barcelona, Spain (Dr. Arturo Evangelista, PI)
* Monaldi Hospital, Naples, Italy (Dr. Giuseppe Limongelli, PI)
* Mayo Clinic, Rochester (Dr. Hector Michelena, PI)
* Oxford University, Oxford, England (Dr. Malenka Bissell, PI)
* San Donato Hospital IRCCS, Milan, Italy (PI: Dr. Alessandro Frigiola)
* Tufts University, Boston (Dr. Gordon Huggins, PI)
* Université Laval, Quebec (Dr. Yohan Bossé, PI)
* University of Michigan, Ann Arbor (Dr. Bo Yang, PI)
* University of Salerno, Salerno, Italy (Dr. Eduardo Bossone, PI)
* University of Texas Medical School, Houston (Dr. Dianna Milewicz, PI) One center with specific expertise, but not enrolling patients, is University of Ottawa (Dr. Mona Nemer, PI).

The data supplied by each participating center are collected from the following sources:

Patient interview or questionnaire Hospital medical records Surgical records Imaging studies

Enrollment Information about the Registry will be disseminated to potential study subjects using a number of sources. The principal means of enrollment will be from the Cardiology and Surgical Clinics of each Hospital. In addition, collaborations with the patient advocacy groups such as the Bicuspid Aortic Valve Foundation. These organizations have well established resources for providing information to patients such as websites, newsletters, and national conferences. A recruitment brochure has been developed to explain the goals and basic procedures of the Registry. Finally, the study website, http://www.bavcon.org, will inform potential subjects about the Registry. All recruitment materials will be approved by the DCC and BCC IRBs, as appropriate, prior to dissemination.

BCC study staff will identify eligible patients using the eligibility criteria developed and approved by the Steering Committee. They will both screen their current patient population as well as identify new patients that attend the clinic. Eligible patients will be solicited during clinic visits according to protocols approved by the local IRB.

Initially, a care provider will introduce the Registry to the patient or the parent or guardian of the patient, and ask if they are interested in talking further with the research coordinator. If the patient (or parent or guardian) agrees, the research coordinator will meet with the patient for a more comprehensive explanation of the Registry. If there is continued agreement, the research coordinator will proceed with the consent and enrollment process. Signed informed consent will be obtained prior to any data or sample collection. Patients will receive a hard-copy of the consent form to keep. Patients will be able to ask questions at any time. One parent or guardian may provide signed consent for a minor child or other person with a physical or mental condition that prevents them from doing so themselves. Literacy in the native language of the country (English and Spanish in the USA) will be required of the consenting patient or parent/guardian. Child assent will be obtained from children at least 8 years of age, or as determined by the local IRB. Across all the sites, we anticipate total enrollment of up to 10,000 patients.

Eligibility Criteria

Inclusion criteria for entry into the Registry are:

* Patients diagnosed with bicuspid aortic valve
* All ages ≥8 years
* Able to provide fully informed consent

Local Site Restrictions Some sites will not be collecting tissue from patients, therefore information on tissue collection will be absent. Some sites do not routinely perform CT or MRI on their patients, so these data will also be absent.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as having a bicuspid aortic valve
* All ages ≥8 years
* Able to provide fully informed consent

Exclusion Criteria:

* None

Ages: 8 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with and without bicuspid aortic valves disease
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2013-11 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Bicuspid aortic valve disease | 10 years
  The first specific aim is to identify the genetic causes of bicuspid aortic valve disease.

SECONDARY OUTCOMES:
The development of thoracic aortic disease in patients with bicuspid aortic valve disease | 10 years
  The second specific aim is to identify genetic and non-genetic factors to cause thoracic aortic disease in BAV patients.

CONTACTS AND LOCATIONS:
Overall Officials: Simon C. Body, MD, MPH, Principal Investigator — Boston University School of Medicine, Anesthesiology Department
Locations (12):
- United States (5):
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Texas Health Science Center at Houston, Houston, Texas
- Laval University, Québec, Quebec, Canada
- Italy (4):
  - Istituto Policlinico San Donato, San Donato Milanese, Milan
  - Monaldi Hospital, Naples
  - Second University of Naples, Naples
  - University of Salerno, Salerno
- Hospital Vall d'Hebron, Barcelona, Spain
- University of Oxford, Oxford, United Kingdom